CLINICAL TRIAL: NCT05963802
Title: Crossover Randomized Controlled Trial to Evaluate the Efficacy and Usability of Artificial Intelligence (ChatGPT) for Health Sciences Students (AIHSS)
Brief Title: Evaluation of the Efficacy and Usability of Artificial Intelligence (ChatGPT) for Health Sciences Students
Acronym: AIHSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carleton University (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Mirella Veras, Principal Investigator, Carleton University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: AIHSS01
Record Dates: First submitted 2023-07-04; First posted 2023-07-27 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Educational Activities; AI (Artificial Intelligence)
Keywords: Artificial intelligence; Education; Health Science Students
MeSH Terms: interventions — Artificial Intelligence; Population Groups

STUDY DESIGN:
Intervention Model Description: We employed a crossover design to ensure equity in the learning experience for all students. This involved assigning students either the ChatGPD (A) or the regular online tools (B) for accessing resources and assisting them with their assignments. During the initial phase of the intervention, participants in group A will utilize ChatGPT to complete their assignments, while participants in Group B will serve as the control group. In the subsequent period, the interventions will switch between the two groups.
Who Masked: Investigator
Masking Description: Participants will be informed about the interventions they will be assigned to, ensuring transparency in the study. However, the investigator responsible for the allocation will be blinded to the group assignment of each participant, maintaining the integrity of the study design. To collect the outcomes, an individual external to the research team will be involved. This approach helps minimize potential bias and ensures the data collection process remains independent and unbiased.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Online tools Group (No Intervention): Group B will serve as the control group in this study. Participants in this group will receive instructions on how to complete the assignment using traditional online tools available on the internet, without the use of artificial intelligence. They will have a timeframe of six days to complete the assignment using these conventional tools. Similar to participants in Arm 1, they will also be required to fill out a survey on technology usability, providing feedback on their experience with the online tools.
- Artificial Intelligence (ChatGPT) Group (Experimental): Participants in Group A will be assigned to utilize ChatGPT as their tool to complete assignments. They will be given a period of six days to utilize artificial intelligence through ChatGPT for assignment completion. Along with the assignment instructions, participants will receive an ethical guideline and specific guidelines on how to effectively utilize ChatGPT. Once the intervention period is concluded, participants will be given a 24-hour window to complete a survey that assesses the usability of the technology. The survey aims to gather valuable feedback on the participants' experience and perception of using ChatGPT for their assignments. In addition, participants in Arm 1 will also be asked to fill out a survey regarding their perception of using artificial intelligence (AI) as an assistance tool to complete their assignments. This survey aims to gather insights into their thoughts, opinions, and attitudes towards utilizing AI in the learning process
  Interventions: Other: Artificial Intelligence (ChatGPT) Group

INTERVENTIONS:
Other: Artificial Intelligence (ChatGPT) Group — Participants in Group A will be assigned to utilize ChatGPT as their tool to complete assignments. They will be given a period of six days to utilize artificial intelligence through ChatGPT for assignment completion. Along with the assignment instructions, participants will receive an ethical guideline and specific guidelines on how to effectively utilize ChatGPT. Once the intervention period is concluded, participants will be given a 24-hour window to complete a survey that assesses the usability of the technology. The survey aims to gather valuable feedback on the participants' experience and perception of using ChatGPT for their assignments. In addition, participants in Arm 1 will also be asked to fill out a survey regarding their perception of using artificial intelligence (AI) as an assistance tool to complete their assignments. This survey aims to gather insights into their thoughts, opinions, and attitudes towards utilizing AI in the learning process.
  Arms: Artificial Intelligence (ChatGPT) Group

SUMMARY:
Crossover Randomized Control trial, in which subjects are randomly assigned to one of two groups: one (ChatGPT) receiving the intervention that is being tested, and the control group receiving usual online resources.

DETAILED DESCRIPTION:
A two-stage randomization strategy will be adopted. The allocation of participants into event groups A and B will be determined through computer-generated randomization in an allocation ratio: 1:1. To address ethical concerns regarding power dynamics between professors and students; the investigators have opted to involve an individual who is independent of the research team. This decision aims to minimize any potential bias or influence that could arise from direct professor involvement in the intervention. This approach helps ensure that the study is conducted fairly and unbiasedly, fostering a research environment that prioritizes equal opportunities for all participants. Both groups will simultaneously work on an assignment (A and B).

The investigators employed a cross-over design to ensure equity in the learning experience for all students. This involved assigning students either the ChatGPD (A) or the regular online tools (B) for accessing resources and assisting them with their assignments. During the initial phase of the intervention, participants in group A will utilize ChatGPT to complete their assignments, while participants in Group B will serve as the control group. In the subsequent period, the interventions will switch between the two groups. To assess the participants' technology usability, both groups will complete pre-and post-questionnaires. Additionally, participants will be requested to fill out a post-intervention questionnaire to evaluate their perceptions of the assistance methods. After a period of a wash-out of 13 days/week, participants who were previously allocated to Group A will be allocated to Group B and the same with participants previously allocated to Group B will be to Group A. This crossover randomized control trial will include 50 health sciences students who are registered to the course Chronic Health Conditions and Disability ( HLTH 3503), Carleton University. During the first part of the intervention, A group will use ChatGPT to complete their assignment, while B participants will act as a control group. In the second week, the interventions will cross over. Both groups' participants will complete a pre-and post-questionnaire to assess their knowledge. Participants will also complete a post-intervention questionnaire to evaluate their perceptions. The System Usability Scale (SUS) will be administered at the end of the interventions and when participants cross over to the other assistance tool. This allows for the assessment of outcomes and comparisons within and between the two intervention arms. By collecting data at multiple points in the study, the investigators can evaluate the effects of each intervention and any potential carryover effects during the crossover period. Additionally, it provides an opportunity to measure changes in outcomes within individual participants as they switch from one intervention to another. The questionnaire about socioeconomic, literacy questions, Benefits of AI and risks and negative experiences associated with AI usage.

ELIGIBILITY:
Inclusion Criteria:

* Health Science students
* Must be registered for the course Chronic Health Conditions and Disability (HLTH 3503), Fall 2023.

Exclusion Criteria:

• Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) scores are 0-100,The average SUS score is 68. | within 24 hours
  Technology usability

SECONDARY OUTCOMES:
Student's perception of artificial intelligence, questionnaire reviwed by experts, No recognised gold standard measurement for outcome. | within 24 hours
  Student's perception about the use of artificial intelligence

CONTACTS AND LOCATIONS:
Overall Officials: Mirella Veras, PhD, Principal Investigator — Carleton University
Locations (1):
- Carleton University, Ottawa, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dwan K, Li T, Altman DG, Elbourne D. CONSORT 2010 statement: extension to randomised crossover trials. BMJ. 2019 Jul 31;366:l4378. doi: 10.1136/bmj.l4378. PMID 31366597
- [Result] Luna A, Casertano L, Timmerberg J, O'Neil M, Machowsky J, Leu CS, Lin J, Fang Z, Douglas W, Agrawal S. Artificial intelligence application versus physical therapist for squat evaluation: a randomized controlled trial. Sci Rep. 2021 Sep 13;11(1):18109. doi: 10.1038/s41598-021-97343-y. PMID 34518568
- [Result] Liu X, Rivera SC, Moher D, Calvert MJ, Denniston AK; SPIRIT-AI and CONSORT-AI Working Group. Reporting guidelines for clinical trial reports for interventions involving artificial intelligence: the CONSORT-AI Extension. BMJ. 2020 Sep 9;370:m3164. doi: 10.1136/bmj.m3164. PMID 32909959
- [Result] Zhou L, Bao J, Setiawan IMA, Saptono A, Parmanto B. The mHealth App Usability Questionnaire (MAUQ): Development and Validation Study. JMIR Mhealth Uhealth. 2019 Apr 11;7(4):e11500. doi: 10.2196/11500. PMID 30973342
- [Derived] Veras M, Dyer JO, Rooney M, Barros Silva PG, Rutherford D, Kairy D. Usability and Efficacy of Artificial Intelligence Chatbots (ChatGPT) for Health Sciences Students: Protocol for a Crossover Randomized Controlled Trial. JMIR Res Protoc. 2023 Nov 24;12:e51873. doi: 10.2196/51873. PMID 37999958